CLINICAL TRIAL: NCT05851417
Title: Investigating a Novel Molecular Imaging Technique, Fast Field-Cycling, for Kidney Health and Disease
Brief Title: Fast Field Cycling Imaging of Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2-095-21
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Kidney Diseases
Keywords: Kidney diseases; Fast Field-Cycling imaging
MeSH Terms: conditions — Kidney Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Live donors (Experimental): Live kidney donors (healthy volunteers).
  Interventions: Device: Fast Field-Cycling (FFC) imaging
- Native kidney damage (Experimental): Patients with native kidney damage (suspected active glomerular or interstitial lesion).
  Interventions: Device: Fast Field-Cycling (FFC) imaging
- Kidney transplants (Experimental): Patients with kidney transplant.
  Interventions: Device: Fast Field-Cycling (FFC) imaging

INTERVENTIONS:
Device: Fast Field-Cycling (FFC) imaging — FFC scan

SUMMARY:
The goal of this pilot study is to explore the utility of Fast Field-Cycling (FFC) imaging in monitoring kidney disease. The main questions it aims to answer are:

* If FFC imaging can differentiate healthy kidney from kidney disease
* If there is an association between FFC imaging and standard clinical tests Participants will provide one blood and on urine sample, and will have one FFC imaging scan.

DETAILED DESCRIPTION:
The kidneys are vital organs responsible for clearance of toxins in the human body. The kidneys age over time and this ageing process is complex, involving changes both to their structure and function, and can be accelerated by disease processes. Without an invasive biopsy procedure, it is often difficult to distinguish between age-related damage from active disease, that could be modified with treatment. Even with a biopsy, certain diseases are often patchy and can be overlooked if missed by the biopsy sample procedure. Alternative imaging approaches have limited ability to differentiate between modifiable and non-modifiable disease processes.

The investigators, based at the University of Aberdeen, have developed a unique magnetic imaging technology, Fast Field-Cycling (FFC) imaging. FFC derives from conventional MRI scanners but has the ability to change its magnetic field strength during a scan. This is equivalent to having many MRI scanners in one device and allows completely new analyses of the behaviour of tissue remodelling to pathological processes, from millimetres to nanometres. This information is invisible to standard MRI scanners and several pilot studies have shown great potential for FFC in cancer and stroke.

This pilot study aims to investigate if FFC can detect changes in kidney microstructure. If FFC imaging shows that it is effective in monitoring kidney disease, then this would contribute to evidence from previous studies promoting the need to develop a new scanner that could be used clinically in the future.

The study will include 20 patients with kidney damage (native or transplant kidneys) and 10 live donors (healthy volunteers). Each participant (patients and live donors) will have urine and blood tests, along with an FFC-MRI scan.

Data analyses will be performed using the appropriate statistical methods depending on the distribution of the variables extracted.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Participants must be aged 18 and above
* Participants who meet the safety criteria for undergoing an MRI scan.
* Participants who can pass through a 50 cm-diameter circular hoop to ensure they will be able to fit inside the scanner
* Participants must be able to give fully informed consent.
* Participants must be mobile enough to be positioned onto the FFC-MRI scanner couch.

Native kidney damage patients:

* Patients referred for a kidney biopsy and laboratory evidence (blood tests and urine abnormalities) of kidney impairment.
* Patients who are newly referred.

Transplant patients:

* Patients with functioning kidney transplant undergoing a kidney biopsy as a part of routine clinical care.
* Patients who are newly referred.

Live donors

• Live kidney donors, patients investigated for potential kidney donation and deemed suitable for donation.

Exclusion Criteria:

Native kidney Damage Patients:

* Patients with single native kidney.
* Patients on dialysis.

Transplant patients:

• Patients with non-functioning kidney transplant.

Live donors

• Live donors who deemed unsuitable for kidney donation by the living kidney donation clinic.

All participants:

* MRI-incompatible conditions, as detected in the MRI safety screening sheet.
* Participants under 18 years old.
* Participants who are unable to give fully informed consent.
* Women who are pregnant.
* Restrictions to mobility that would prevent the correct positioning in the scanner.
* Participants who suffer from claustrophobia.
* Body mass index larger than 34, due to the limited bore size of the scanner.
* Participants who are unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Kidney microstructure assessed by Fast Field Cycling (FFC) imaging scan | At baseline
  Evaluating the potential of FFC T1 dispersion profiles in the clinical assessment of kidney microstructure

CONTACTS AND LOCATIONS:
Overall Officials: Simon Sawhney, Dr, Study Chair — NHS Grampian
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No